CLINICAL TRIAL: NCT05419323
Title: Improving Access to Sleep Apnea Care: A Pragmatic Study of New Consultation Models
Brief Title: Direct Referral for Apnea Monitoring
Acronym: DREAM
Status: Active, not recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IIR 15-339; 19-27 (Other: San Francisco Veterans Affairs Medical Center)
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: sleep apnea syndromes; polysomnography; home sleep apnea testing
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Traditional clinical pathway for OSA: After referral, patients will have an initial encounter with a sleep care provider which might include in-person visits, telephone clinics, or video conferencing.
  Intervention/Treatment: Patients in Arm 1 will receive routine care for OSA at one of the participating VA Sleep Medicine clinics.
- DREAM clinical pathway for OSA: After referral, patients will not have an initial encounter with a care provider. After a clinician conducts a chart review of medical records, patients in the DREAM pathway will be referred for sleep testing.
  Intervention/Treatment: Patients in Arm 2 will receive routine care for OSA at one of the participating VA Sleep Medicine clinics.
- Negative predictive value of HSAT: Results of sleep tests will be compared for patients who undergo both HSAT and polysomnographic (PSG) procedures.
  Intervention/Treatment: Patients in Arm 3 will undergo
  a) HSAT sleep testing followed by PSG testing, or b) simultaneous administration of PSG and HSAT sleep testing.

SUMMARY:
The primary objective of this project is to compare a health care delivery model, Direct Referral for Apnea Monitoring (DREAM), with initial in-person (Traditional) clinic appointments for Veterans at risk for obstructive sleep apnea (OSA). A secondary objective is to determine the negative predictive value (NPV) of home sleep apnea testing (HSAT).

DETAILED DESCRIPTION:
Patients referred to one of 3 participating VA sleep medicine clinics (San Francisco VA, VA Portland or VA Pittsburgh) for OSA will be assigned either to the Traditional clinical pathway (which might include an initial encounter with a sleep care provider through in-person visits, telephone clinics, or video conferencing) or the DREAM pathway which will omit the initial encounter with a care provider. After a clinician conducts a chart review of medical records, patients in the DREAM pathway will be referred for sleep testing. All patients will be tracked from the time of referral until 90-days past the initiation of treatment. To determine the NPV of HSAT, results of sleep tests will be compared for patients who undergo both HSAT and polysomnographic (PSG) procedures. Concurrent PSG and HSAT studies will be done at Portland, Pittsburgh, and San Francisco.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years Agrees to be seen by a VA sleep program Reason for referral to sleep clinic: New OSA Evaluation

Exclusion Criteria:

Age < 18 years Declines to be seen by a VA sleep program Reason for referral to sleep clinic: anything other than a new OSA evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will include patients referred for new OSA evaluations at Sleep Medicine clinics at the 3 VA study sites. Participants will be identified via a review of their medical records by the PIs (study physicians) after they are referred for OSA evaluations at the 3 study sites.
Sampling Method: Non-Probability Sample
Enrollment: 6501 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Time from referral | 1 year
  For Arms 1 & 2: Compare time from referral to sleep testing and treatment of OSA
PAP adherence | 1 year
  For Arms 1 & 2: PAP treatment adherence (for example, Percentage of days with usage >= 4 hours) between Traditional and DREAM clinical pathways
AHI scores | 4 years
  For Arm 3: Compare apnea-hypopnea index (AHI) scores between HSAT and PSG procedures

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Fumiko Sarmiento, MD MPH, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (3):
- United States (3):
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared at the conclusion of this study.
Supporting Information: Study Protocol, SAP
Time Frame: From study initiation to completion, 2020-2025

REFERENCES:
- [Background] Folmer RL, Smith CJ, Boudreau EA, Hickok AW, Totten AM, Kaul B, Stepnowsky CJ, Whooley MA, Sarmiento KF. Prevalence and management of sleep disorders in the Veterans Health Administration. Sleep Med Rev. 2020 Dec;54:101358. doi: 10.1016/j.smrv.2020.101358. Epub 2020 Jul 20. PMID 32791487
- [Background] Sarmiento KF, Boudreau EA, Smith CJ, Kaul B, Johnson N, Folmer RL. Effects of Computer-Based Documentation Procedures on Health Care Workload Assessment and Resource Allocation: An Example From VA Sleep Medicine Programs. Fed Pract. 2020 Aug;37(8):368-374. doi: 10.12788/fp.0023. PMID 32908344
- [Background] Chang YHA, Folmer RL, Shasha B, Shea JA, Sarmiento K, Stepnowsky CJ, Lim D, Pack A, Kuna ST. Barriers and facilitators to the implementation of a novel web-based sleep apnea management platform. Sleep. 2021 Apr 9;44(4):zsaa243. doi: 10.1093/sleep/zsaa243. PMID 33216916
- [Background] Atwood CW, Boudreau EA, Folmer RL, Kuna ST, Pineda L, Reichert J, Sarmiento K, Thompson W, Whooley M, Zhang N, Yarbrough WC. 1170 Trends in Sleep Apnea Testing Among Veterans Participating in a Rural Health-Focused Telesleep Medicine Program. [Abstract]. Sleep Medicine Reviews. 2020 Apr 1; 43(Supplement 1):A447.
- [Background] Salinsky M, Evrard C, Joos S, Boudreau E. Utility of mental health and sleep screening questionnaires for patients admitted to a seizure monitoring unit. Epilepsy Behav. 2021 Oct;123:108237. doi: 10.1016/j.yebeh.2021.108237. Epub 2021 Aug 7. PMID 34375800
- [Background] Sarmiento K, Kuna S, Boudreau EA, Atwood C, Pineda L, Thompson W, Zeidler M, Fields B, Uzzaman A, Totten A, Smith C, Folmer RL, Williams K, Zhang N, Whooley M. VHA's TeleSleep Program improves rural Veteran access to sleep care through expansion of telehealth networks. [Abstract]. Sleep. 2021 May 3; 44(Suppl 2):A317-A318.
- [Background] Folmer RL, Boudreau EA, Atwood CW, Smith CJ, Totten AM, Tock JL, Chilakamarri P, Sarmiento KF. Study protocol to assess de-implementation of the initial provider encounter for diagnosis and treatment of obstructive sleep apnea: the DREAM (Direct Referral for Apnea Monitoring) Project. BMC Pulm Med. 2022 Apr 2;22(1):123. doi: 10.1186/s12890-022-01899-y. PMID 35366836
- [Background] Atwood W, Smith C, Totten A, Boudreau EA, Sarmiento K, Hahn Z, Folmer RL, Tock J, Hotchkiss J. Good Sleep Care: Geospatial Optimization of Distant Sleep Care in the VA. [Abstract]. Sleep. 2022 Jun 1; 45(Suppl 1):A164.
- [Result] Folmer RL, Smith CJ, Boudreau EA, Totten AM, Chilakamarri P, Atwood CW, Sarmiento KF. Sleep disorders among rural Veterans: Relative prevalence, comorbidities, and comparisons with urban Veterans. J Rural Health. 2023 Jun;39(3):582-594. doi: 10.1111/jrh.12722. Epub 2022 Nov 5. PMID 36333991
- [Result] Chun VS, Whooley MA, Williams K, Zhang N, Zeidler MR, Atwood CW, Folmer RL, Totten AM, Smith CJ, Boudreau EA, Reichert JM, Sarmiento KF. Veterans Health Administration TeleSleep Enterprise-Wide Initiative 2017-2020: bringing sleep care to our nation's veterans. J Clin Sleep Med. 2023 May 1;19(5):913-923. doi: 10.5664/jcsm.10488. PMID 36708262
- [Result] Hahn Z, Hotchkiss J, Atwood C, Smith C, Totten A, Boudreau E, Folmer R, Chilakamarri P, Whooley M, Sarmiento K. Travel Burden as a Measure of Healthcare Access and the Impact of Telehealth within the Veterans Health Administration. J Gen Intern Med. 2023 Jul;38(Suppl 3):805-813. doi: 10.1007/s11606-023-08125-3. Epub 2023 Jun 20. PMID 37340257
- [Result] Folmer RL. Unresolved Issues Associated with Transcranial Magnetic Stimulation (TMS) Treatment of Chronic Tinnitus. J Clin Med. 2023 Jul 12;12(14):4648. doi: 10.3390/jcm12144648. PMID 37510763
- [Result] Mazzotti DR, Haendel MA, McMurry JA, Smith CJ, Buysse DJ, Roenneberg T, Penzel T, Purcell S, Redline S, Zhang Y, Merikangas KR, Menetski JP, Mullington J, Boudreau E. Sleep and circadian informatics data harmonization: a workshop report from the Sleep Research Society and Sleep Research Network. Sleep. 2022 Jun 13;45(6):zsac002. doi: 10.1093/sleep/zsac002. PMID 35030631
- [Result] Belkora JK, Ortiz DeBoque L, Folmer RL, Totten AM, Williams K, Whooley MA, Boudreau E, Atwood CW, Zeidler M, Rezayat T, Chilakamarri P, Sarmiento KF. Sustainment of the TeleSleep program for rural veterans. Front Health Serv. 2023 Nov 10;3:1214071. doi: 10.3389/frhs.2023.1214071. eCollection 2023. PMID 38028943
- [Result] Atwood C, Boudreau EA, Sarmiento K, Williams K, Totten A, Folmer RL, Wholey M. 1058 Experience of VA Telesleep Medicine Following the COVID Pandemic. [Abstract]. Sleep. 2024 May 1; 47(Suppl 1):A454-A455.
- [Result] Shamim-Uzzaman QA, Zeidler MR, Boudreau EA, Chowdhuri S, Donovan LM, El-Solh A, Freire AX, Gottlieb DJ, Jindal RD, Hesselbacher S, Koo B, Kuna S, Lim MM, Mina S, Stepnowsky C, Tamanna S, Tobias L, Ulmer C, Yaggi K, Surani S, Atwood C, Sarmiento K, Ioachimescu OC. Sleep research, quality and implementation priorities in the Veterans Health Administration: a white paper. J Clin Sleep Med. 2025 Oct 1;21(10):1787-1797. doi: 10.5664/jcsm.11734. PMID 40375810